CLINICAL TRIAL: NCT02498782
Title: Phase 2, Randomized, Multicenter, Placebo-controlled, Safety and Efficacy Study to Evaluate Six Oral Fexinidazole Dosing Regimens for the Treatment of Adult Patients With Chronic Indeterminate Chagas Disease.
Brief Title: Study to Evaluate Fexinidazole Dosing Regimens for the Treatment of Adult Patients With Chagas Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNDi-CH-FEXI-001
Record Dates: First submitted 2014-08-20; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Chagas Disease; Trypanosomiasis, South American; South American Trypanosomiasis; Disease, Chagas
Keywords: Chagas Disease; Dosage forms; Regimens
MeSH Terms: conditions — Chagas Disease | interventions — fexinidazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Fexinidazole, 1800 mg, 2 weeks (Active Comparator): 1800mg (High Dose) 2 weeks (HD - 2 weeks) Group: Fexinidazole, 1800 mg QD for 2 weeks, followed by placebo to complete 8 weeks (total dose: 25,2 g)
  Interventions: Drug: Fexinidazole; Drug: Placebo
- Fexinidazole, 1800 mg, 4 weeks (Active Comparator): 1800mg (High Dose) 4 weeks (HD - 4 weeks) Group: Fexinidazole, 1800 mg QD for 4 weeks, followed by placebo to complete 8 weeks (total dose: 50,4 g)
  Interventions: Drug: Fexinidazole; Drug: Placebo
- Fexinidazole, 1800 mg, 8 weeks (Active Comparator): 1800mg (High Dose) 8 weeks (HD - 8 weeks) Group: Fexinidazole, 1800 mg QD, for 8 weeks (total dose: 100,8 g)
  Interventions: Drug: Fexinidazole
- Fexinidazole, 1200 mg, 2 weeks (Active Comparator): 1200mg (Dose 2 weeks) 2 weeks (LD - 2 weeks) Group: Fexinidazole, 1200 mg QD for 2 weeks, followed by placebo to complete 8 weeks (total dose: 16,8 g)
  Interventions: Drug: Fexinidazole; Drug: Placebo
- Fexinidazole, 1200 mg, 4 weeks (Active Comparator): 1200mg (Low Dose) 4 weeks (LD - 4 weeks) Group: Fexinidazole, 1200 mg QD for 4 weeks, followed by placebo to complete 8 weeks (total dose: 33,6 g)
  Interventions: Drug: Fexinidazole; Drug: Placebo
- Fexinidazole, 1200 mg, 8 weeks (Active Comparator): 1200mg (Low Dose) 8 weeks (LD - 8 weeks) Group: Fexinidazole, 1200 mg QD for 8 weeks (total dose: 67,2 g)
  Interventions: Drug: Fexinidazole
- Placebo (Placebo Comparator): Placebo (8 weeks) Group: Fexinidazole matched placebo tablets QD for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fexinidazole
  Other Names: 1Himidazole,1methyl2[4methylthio)phenoxymethyl] 5nitroimidazole
  Arms: Fexinidazole, 1200 mg, 2 weeks; Fexinidazole, 1200 mg, 4 weeks; Fexinidazole, 1200 mg, 8 weeks; Fexinidazole, 1800 mg, 2 weeks; Fexinidazole, 1800 mg, 4 weeks; Fexinidazole, 1800 mg, 8 weeks
Drug: Placebo
  Arms: Fexinidazole, 1200 mg, 2 weeks; Fexinidazole, 1200 mg, 4 weeks; Fexinidazole, 1800 mg, 2 weeks; Fexinidazole, 1800 mg, 4 weeks; Placebo

SUMMARY:
The hypothesis is to evaluate if the treatment with Fexinidazole will lead to a better sustained clearance of the parasites at 6 months of follow-up when in comparison to placebo in patients with chronic indeterminate CD.

DETAILED DESCRIPTION:
Chagas Disease (CD) ranks among the world's most neglected diseases. In Latin America, 21 countries are endemic for CD with an estimated 100 million people at risk of contracting the disease. Estimates from the 1980s indicated that some 16 million to 18 million individuals were infected. In the 1990s, after a series of multinational control initiatives, estimates of the number of infected people were revised to 9.8 million in 2001. The estimated burden of disease in terms of disability-adjusted life years (DALYs) declined from 2.7 million in 1990 to 586,000 in 2001. Recent estimates from PAHO (2006) indicate 7.54 million infected people and 55,185 new cases per year. New safe and effective treatments for Chagas Disease are urgently needed. Current chemotherapy options for CD have significant limitations, including long treatment durations, and safety and tolerability concerns. For many years, inhibitors of the sterol biosynthesis pathway, such as posaconazole and ravuconazole, were considered as the most promising new drugs candidates for Chagas Disease. Following the recent results of CHAGAZASOL, an investigator-initiated trial conducted in Barcelona, where a high recrudescence rate was observed in the posaconazole treatment arms (80-90%, versus 5% in the benznidazole arm), there is increased concern on the future of the class. Nitroimidazoles are a well-known class of pharmacologically active compounds, among which several have shown good activity against trypanosomes. While concerns over mutagenicity and safety have mitigated their potential as drug candidates, several members of this family are widely used as antibiotics, indicating that it is possible to select compounds with acceptable activity/toxicity profile in this class. Fexinidazole had been in preclinical development as a broad-spectrum antiprotozoal drug by Hoechst in the 1970s-1980s, but its clinical development was not pursued at the time. The molecule was ''rediscovered'' and selected for development by the Drugs for Neglected Diseases initiative (DNDi) as a new drug candidate for sleeping sickness, following a systematic review and profiling of more than 700 nitroheterocyclic compounds (mostly nitroimidazoles) from diverse sources, which included assessments of antiparasitic activity and mutagenic potential. Fexinidazole underwent extensive regulatory toxicology studies, including safety pharmacology (respiratory, cardiovascular, and general behaviour) and 4 weeks of repeated dose toxicokinetics studies in rat and dogs. 90-day toxicology studies were performed by Hoechst, allowing validation of the 3 months dosing in rat to a dose of 800 mg/kg/day and dog up to 125 mg/kg/day. Overall, Fexinidazole was found to be well tolerated, with no specific toxicity or other concerns.

During 2010-2011, DNDi carried out several Phase I clinical trials assessing the safety and pharmacokinetics of Fexinidazole in human volunteers given in single and multiple doses. A pivotal phase II/III clinical safety and efficacy study in sleeping sickness patients was started in 2012 and to-date shows encouraging safety and tolerability profile and exposure in patients.

Fexinidazole has previously been described as effective and superior to benznidazole or nifurtimox in one acute murine infection model with the T. cruzi Brazil 32 strain, but the methodologies used to establish cure are no longer considered the most accurate. More recently, in vitro studies performed at Institute Pasteur Korea (IPK) showed that Fexinidazole parent and metabolites (M1 and M2) are more or less equipotent versus T. cruzi in vitro (Tulahuen strain). Fexinidazole Sulfone (M2) is potent against a panel of T. cruzi strains (not including Colombiana or VL-10) albeit at higher concentrations than Benznidazole (2 to 4-fold). Fexinidazole Sulfone requires 72 to 96 hrs exposure at concentrations at or above 100 mM (31 mg/ml) with the Y strain; Benznidazole exhibits the same kinetics but requires exposure at the lower concentration of 12.5 mM (3.3 mg/ml).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of T. cruzi infection by Serial qualitative PCR (three samples collected over a single day, at least one of which must be positive) AND Conventional serology (a minimum of two out of three positive tests must be positive [Conventional ELISA, Recombinant Elisa or IIF)
* Women in reproductive age must have a negative serum pregnancy test at screening, must not be breastfeeding, and consistently use a highly effective contraceptive method during the entire trial.
* Normal EKG (PR ≤200 msec, QRS ≤120 msec, and QTc ≥400msec and ≤450 msec interval durations) at screening

Exclusion Criteria:

* Signs and/or symptoms of chronic cardiac and/or digestive form of CD (as per Study Manual of Operations)
* History of cardiomyopathy, heart failure or ventricular arrhythmia
* Any other acute or chronic health conditions that, in the opinion of the PI, may interfere with the efficacy and/or safety evaluation of the study drug (such as acute infections, history of HIV infection, diabetes, liver and renal disease requiring medical treatment)
* Laboratory test values considered clinically significant or out of the allowable range at screening as follows:

  * Total WBC must be within the normal range, with an acceptable margin of +/- 5% (3,800 - 10,500 / mm3).
  * Platelets must be within the normal range up to 550,000 / mm3
  * Total bilirubin must be within the normal range Transaminases (ALT and AST) must be within the normal range, with an acceptable margin of 25% above the upper limit of normality (ULN), < 1.25 x ULN.
  * Creatinine must be within an acceptable margin of 10% above the ULN, <1.10 x ULN.
  * Alkaline phosphatase must be within the normal range up to Grade 1 CTCAE (< 2.5 x ULN)
  * GGT must be within the normal range up to 2x ULN.
  * Potassium, Magnesium, Calcium must be within the normal range
* History of alcohol abuse or any other drug addiction (as specified in the Study Manual of Operations).
* Any condition that prevents the patient from taking oral medication.
* Patients with contra-indication (known hypersensitivity) to other nitroimidazoles, e.g. metronidazole.
* Any concomitant use of antimicrobial or anti-parasitic agents.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-09 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Parasitological cure rate (PCR) | 8 weeks and sustained until 6 months
  Parasitological cure rate as determined by serial negative qualitative PCR results (3 negative PCR results, from 3 samples to be collected in the same day) at end of treatment (8 weeks) and sustained parasitological clearance until 6 months follow-up.
Adverse events | 7 months
  Incidence and severity of adverse events (clinical, laboratory and EKG)
Serious Adverse events | 7 months
  Incidence of Serious Adverse Events and/or adverse events leading to treatment discontinuation

SECONDARY OUTCOMES:
Parasite Clearance (qualitative PCR) | weeks 2, 3, 4, 6, 10, and at 4 and 6 months follow-up
  Parasite clearance at weeks 2, 3, 4, 6, 10, and at 4 and 6 months follow-up as measured by qualitative PCR
Parasite load | weeks 2, 3, 4, 6, 10 and 4 and 6 months
  Change in parasite load over time assessed at weeks 2, 3, 4, 6, 10, and at 4 and 6 months follow-up as measured by quantitative PCR
Serological response | week 10, 4 and 6 months
  Serological response (conventional and non-conventional serologies) (incidence of conversion to negative and changes in titers over time) assessed at week 10 and at 4 and 6 months follow-up.
Blood culture for parasite genotyping | 6 months
  Blood culture and in vitro drug and susceptibility testing of isolated parasite strains at 6 months.

OTHER OUTCOMES:
Plasma level concentrations | D0 (pre-dose), at randomly selected time at day 1, post-dose, at steady-state phase (week 2-9), and at week 10
  Plasma level concentrations of Fexinidazole and its metabolites M1 (sulfoxide) and M2 (sulfone) will be determined at D0 (pre-dose), at randomly selected time after first day of treatment administration (day 1, post-dose), at steady-state phase (week 2-9), and at week 10

CONTACTS AND LOCATIONS:
Overall Officials: Faustino Torrico, MD, Principal Investigator — Plataforma de Antención Integral de Pacientes con Enfermedad de Chagas, Cochabamba, Bolivia; Joaquim Gascón, MD, Principal Investigator — Centro de Salud Internacional, Hospital Clínico de Barcelona; Lourdes O Daza, MD, Principal Investigator — Plataforma de Antención Integral de Pacientes con Enfermedad de Chagas, Tarija, Bolivia
Locations (2):
- Bolivia (2):
  - Plataforma Atención Integral de Pacientes con Enfermedad de Chagas, Cochabamba
  - Plataforma de Atención Integral de Pacientes con Enfermedad de Chagas, Tarija

REFERENCES:
- [Derived] Torrico F, Gascon J, Ortiz L, Pinto J, Rojas G, Palacios A, Barreira F, Blum B, Schijman AG, Vaillant M, Strub-Wourgaft N, Pinazo MJ, Bilbe G, Ribeiro I. A Phase 2, Randomized, Multicenter, Placebo-Controlled, Proof-of-Concept Trial of Oral Fexinidazole in Adults With Chronic Indeterminate Chagas Disease. Clin Infect Dis. 2023 Feb 8;76(3):e1186-e1194. doi: 10.1093/cid/ciac579. PMID 35925555